CLINICAL TRIAL: NCT03406377
Title: A Phase 2, Double-blind Dose Escalation Regimen of Once-Weekly OPK-88003 in Subjects With Type 2 Diabetes
Brief Title: Effects and Safety of OPK-88003 Dose Escalation in Type 2 Diabetes Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DPO-203
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Water for injection, Sorbitol, L-Methionine, Sodium Acetate Trihydrate
  Interventions: Drug: Placebo
- OPK-88003 (Experimental): 70 mg/vial (extractable volume 1 mL) (20mg for 4 weeks, 40 mg for 4 weeks and 70 mg for 22 weeks)
  Interventions: Drug: OPK-88003

INTERVENTIONS:
Drug: OPK-88003 — OPK-88003 subcutaneous injection
  Arms: OPK-88003
Drug: Placebo — Placebo subcutaneous injection
  Arms: Placebo

SUMMARY:
This study will evaluate the effect of dose escalation of once-weekly (QW) subcutaneous (SC) OPK-8003 injections vs placebo on HbA1c absolute change from baseline at 30 weeks in subjects with type 2 diabetes mellitus (T2DM) inadequately controlled with diet and exercise alone, or treated with a stable dose of metformin.

DETAILED DESCRIPTION:
This clinical trial is a phase 2, double-blind dose escalation regimen of once-weekly OPK-88003 in subjects with T2DM. The trial consists of a screening/baseline (up to 2 weeks prior to first dose), treatment period consisting of a dose escalation (8 weeks) and a target dose (22 weeks), and a follow-up period (4 weeks). Subjects will be randomly assigned to volume-matched OPK-88003 or placebo administered QW.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 to 80 years with T2DM treated with diet and exercise alone or on a stable dose of metformin (≥ 1000 mg/day),
* BMI ≥27 and ≤45 kg/m2
* HbA1c ≥7.0% and ≤10.5% at screening

Exclusion Criteria:

* Type 1 diabetes mellitus
* Previous treatment with incretin mimetic drugs
* Have used insulin for diabetic control for more than 6 consecutive days within the prior year
* Have had two or more emergency room visits or hospitalizations due to poor glucose control within the prior 6 months
* Have a history of acute or chronic pancreatitis or elevation in serum lipase/amylase (>2 x ULN).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Militza Vera De Alba, MD, Study Director — OPKO Health, Inc.
Locations (3):
- United States (3):
  - National Research Institute - Huntington Park, Huntington Park, California
  - National Research Institute - Wilshire, Los Angeles, California
  - Clinical Pharmacology of Miami, LLC, Hialeah, Florida

RESULTS

PARTICIPANT FLOW:
Groups:
- OPK-88003: 70 mg/vial (extractable volume 1 mL)
  OPK-88003: OPK-88003 subcutaneous injection
Period: Overall Study
Arm/Group | Placebo | OPK-88003
Started | 41 | 72
Completed | 25 | 51
Not Completed | 16 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | OPK-88003 | Total
Number analyzed (Participants) | 41 | 72 | 113
Age, Continuous [Mean (Standard Deviation); unit: Year] | 57.4 (9.06) | 53.8 (9.94) | 55.1 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 29 | 53
  Male | 17 | 43 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 36 | 59
  Not Hispanic or Latino | 18 | 36 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 12 | 18
  White | 33 | 60 | 93
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c in Subjects With Type 2 DM
Description: To evaluate the effect of dose escalation of QW SC OPK-88003 vs placebo injections on HbA1c absolute change from baseline to after 30 weeks treatment in subjects with T2DM inadequately controlled with diet and exercise alone, or treated with a stable dose of metformin.
Time Frame: From baseline to 30 weeks
Measure: Least Squares Mean (Standard Error); unit: mmols/mol
Arm/Group | Placebo | OPK-88003
Number analyzed (Participants) | 28 | 45
mmols/mol | -0.25 (0.209) | -1.47 (0.168)

2. Secondary Outcome: Mean Percent (%) Body Weight Change
Description: Mean percent (%) body weight change from baseline to after 30 weeks treatment
Time Frame: From baseline to 30 weeks
Measure: Least Squares Mean (Standard Error); unit: Percentage of body weight change
Arm/Group | Placebo | OPK-88003
Number analyzed (Participants) | 28 | 45
Percentage of body weight change | -2.10 (0.976) | -5.83 (0.737)

3. Secondary Outcome: Percent (%) of Subjects With 5% or Greater Body Weight Loss.
Description: Percent (%) of subjects with 5% or greater body weight loss after 30 weeks treatment
Time Frame: 30 weeks.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | OPK-88003
Number analyzed (Participants) | 28 | 45
Percentage of participants | 16.7 | 48.8

4. Secondary Outcome: Change From Baseline of Fasting Plasma Glucose (FPG).
Description: Change of FPG from baseline to after 30 weeks treatment
Time Frame: 30 weeks.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | OPK-88003
Number analyzed (Participants) | 28 | 45
mg/dL | -13.3 (7.04) | -46.2 (5.86)

ADVERSE EVENTS:
Time Frame: 36 weeks
Arm/Group | Placebo | OPK-88003
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/72
Serious Adverse Events (participants affected / at risk) | 2/41 | 9/72
Other Adverse Events (participants affected / at risk) | 5/41 | 35/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | OPK-88003 (N=72)
Branch retinal artery occlusion (Eye disorders) | 0 | 1
Branch retinal artery occlusion account for peripheral vision loss right eye (Eye disorders) | 0 | 1
Acute cholelithiasis (Hepatobiliary disorders) | 0 | 1
Acute pancreatitis (Gastrointestinal disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Hypersensitivity reaction (Immune system disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Renal calculi (Renal and urinary disorders) | 0 | 1
Right fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Right distal tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Small bowel obstruction (Gastrointestinal disorders) | 0 | 1
Non st-segment elevation myocardial infarction (Cardiac disorders) | 0 | 1
Acute diverticulitis (Infections and infestations) | 0 | 1
Cecal volvulus s/p right hemicolectomy (Gastrointestinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Acute toxic encephalopathy (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | OPK-88003 (N=72)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 28
Vomiting (Gastrointestinal disorders) | 1 | 19
Diarrhoea (Gastrointestinal disorders) | 3 | 9
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Lipase increased (Investigations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT03406377/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT03406377/SAP_001.pdf